CLINICAL TRIAL: NCT00512239
Title: Early Prediction of Patient-related and Radiological Outcomes in Patients With Recent-onset Inflammatory Polyarthritis (EPA) Using Established and Novel Independent Predictors
Brief Title: Prognostic Evaluation of Inflammatory Polyarthritis of Recent Onset
Acronym: EUPA
Status: Recruiting | Type: Observational
Sponsor: Gilles Boire (Other)
Collaborators: The Arthritis Society, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Gilles Boire, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: EUPA97-04; CIHR MOP-110959 (Other Grant/Funding Number: Canadian Institutes for Health Research)
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis
Keywords: Early Rheumatoid Arthritis; Early inflammatory arthritis; Biomarkers; Autoantibodies; Anti-Sa antibodies; Anti-CCP antibodies
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, genomic DNA and RNA from peripheral blood, peripheral blood mononuclear cells (PBMCs) used for in vitro osteoclastogenesis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EUPA cohort: Consecutive adult patients presenting to receive rheumatological care at the Sherbrooke University Hospital Centre (CHUS) with an immune-mediated inflammatory arthritis affecting at least 3 joints for a duration of more than 4 and less than 52 weeks.

SUMMARY:
Inflammatory joint diseases are major causes of invalidity and morbidity. Rheumatoid arthritis (RA), the most frequent of chronic arthritides, affects close to 1% of the Canadian population. Direct and indirect costs of RA represent close to 1% of the gross national product. Recent evidence suggest that initiation of early (e.g., during the first 3-12 months of disease) aggressive treatment decreases both mortality and long term invalidity in RA and other chronic arthritides. However, a significant proportion of patients with early polyarthritis (EPA) have a benign evolution, even if they fulfill criteria for RA. On the contrary, most patients whose arthritis persist for more than 12 months have a progressive and destructive disease. Currently available clinical, serological and genetic markers of severity in arthritic patients perform poorly in EPA patients to identify those patients whose arthritis is likely to persist and thus who deserve an aggressive treatment.

The Investigators propose a prospective and longitudinal study to define the contribution of detection of rheumatoid arthritis-specific autoantibodies (RASA), either alone or in combination with other markers of severity, in the prognostic evaluation of patients presenting with EPA. Availability of such an effective serological tool to establish prognosis in individual patients would improve therapeutic decisions in clinical practice. The same prognostic tools would represent very powerful instruments to subset patients into more homogeneous groups in clinical trials, increasing their power.

DETAILED DESCRIPTION:
Inflammatory polyarthritides are major causes of invalidity and morbidity. Treatment of rheumatoid arthritis (RA), the most common and most severe of these diseases, is clearly more effective when initiated early using aggressive therapeutic protocols. The recent availability of very effective but extremely costly biologic agents may further improve our treatment strategies. Specific arthritides (e.g., RA) were defined using sets of criteria that are unable to define prognosis and cannot be used to select which patients, early in the course of their disease, should be treated aggressively. A number of putative prognostic markers of severity are available, including anti-Sa and anti-Cyclic Citrullinated peptides (Anti-CCP) antibodies (Abs), whose presence is highly specific to RA. Anti-Cit Abs might characterize one of the severe subsets of RA, both clinically and pathogenically. However, these markers are not yet demonstrated to risk-stratify patients with arthritis of recent onset.

Objectives. Our PRIMARY objectives are to evaluate the sensitivity, specificity, and positive likelihood ratios (+LR) of anti-Sa Abs to identify among patients with early polyarthritis (EPA) in the first 12 months of disease (median 4 months) those that will, at 18, 30, 42 and 60 months into disease : 1- have persistent arthritis; 2- satisfy American College of Rheumatology (ACR) criteria for RA; 3- have developed a SEVERE disease (as defined by their Sharp/van der Heijde radiological score or their modified Health Assessment Questionnaire (M-HAQ) score, as well as by our composite index that includes both scores).

In particular, we want to evaluate the size of the ADDITIONAL independent contribution of anti-Sa Abs to predict severe disease, when added to markers of poor prognosis in established RA (e.g., immunoglobulin M (IgM) Rheumatoid Factor (RF), "shared epitope", persistent high C-Reactive Protein (CRP) levels).

Our SECONDARY objectives are to evaluate the sensitivity, specificity, and +LR : 1- of anti-CCP and anti-Sa Abs (individually and in sets) to identify among patients with EPA those who will develop a SEVERE disease after 18, 30, 42, and 60 months; 2- of novel genetic markers to identify among patients with EPA those that will develop a SEVERE disease after 18, 30, 42, and 60 months; 3- of anti-Sa and anti-CCP Abs to identify among patients with EPA those patients who will require more intensive anti-rheumatic treatment (DMARD combinations and/or biologics) at 18, 30, 42 and 60 months; and 4- of serum and urine markers of cartilage degradation and regeneration to identify among patients with EPA those that will develop a SEVERE disease after 18, 30, 42, and 60 months.

Methods. We set up a single-center longitudinal observational study (LOS) planned to include 390 consecutive EPA patients observed over 5 years. EPA is defined as synovitis affecting 3 or more joints for more than one month and less than 12 months, with few specific exclusions. At inclusion, and at each pre-defined time points after disease onset, extensive (but focused) demographic, clinical, serological, radiological and genetic data are collected, without interference with their treatment. Treating physicians and patients remain uninformed about the status of the patients regarding research data (genomic data, anti-Sa and anti-CCP Abs). About 250 such patients will have been included at the time of renewal. Loss to follow up (up to V4 in some patients) at each visit is about 5% and is mostly found in patients in remission. Data collected are used to verify whether patients have reached predefined outcomes including remission, persistence of arthritis, persistence of arthritis fulfilling RA criteria, DMARD use, and SEVERE disease.

Discussion. We have now assembled a large cohort of patients with EPA that are thoroughly reassessed at regular intervals, allowing stratification of patients using outcome measures that have been set in advance. The information gained from this study may have very significant therapeutic and economic implications.

ELIGIBILITY:
Inclusion Criteria:

* Early Rheumatoid arthritis
* Early Inflammatory Arthritis

Exclusion Criteria:

* Refusal or inability to consent
* Infectious arthritis
* Microcrystalline arthritis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent-onset inflammatory polyarthritis with an immune cause (excluding infection, crystal-induced) and without characteristics diagnostic for connective tissue diseases or systemic vasculatidies
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1998-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Role of anti-Sa antibodies as predictor of severe radiographical damage | At 60 months after symptom onset
  Proportion of patients who have detectable damage (that is a score of least 5, the minimally detectable difference) on radiographs of hands, wrists and feet according to Sharp score modified by van der Heijde (0-448; higher scores indicative of more damage)

SECONDARY OUTCOMES:
Role of anti-Sa antibodies as predictor of the use of advanced therapy | At baseline and annually over 60 months after symptom onst
  Proportion of patients who use advanced therapies (biologics and Jak inhibitors) at the time of the visit
Role of anti-Sa antibodies as predictor of persistent disease activity | At inclusion and annually over 60 months after symptom onset
  Proportion of patients who fail to reach remission in disease activity at the time of the visit according to Simple Disease Activity Index (SDAI; 0.1-96; a higher score means higher disease activity; a score below 3.3 indicates remission)
Role of psychosocial determinants as predictors of severe outcomes | At baseline and annually over 60 months after symptom onset
  Proportion of participants who fail to reach remission at the time of the visit according to Simple Disease Activity Index (SDAI)

OTHER OUTCOMES:
Epigenetic predictors of severe outcomes | At baseline and annually over 60 months from symptom onset
  Proportion of patients who have detectable damage (that is a score of least 5, the minimally detectable difference) on radiographs of hands, wrists and feet according to Sharp score modified by van der Heijde (0-448; higher scores indicative of more damage)
Epigenetic predictors of persistent disease activity | At baseline and annually over 60 months after symptom onset
  Proportion of participants who fail to reach remission at the time of the visit according to Simple Disease Activity Index (SDAI)
Genetic predictors of severe outcomes | At baseline and annually over 60 months after symptom onset
  Proportion of patients who have detectable damage (that is a score of at least 5, the minimally detectable difference) on radiographs of hands, wrists and feet according to Sharp score modified by van der Heijde (0-448; higher scores indicative of more damage)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD, MSc, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Anonymized data to be shared following individual agreements

REFERENCES:
- [Background] Maksymowych WP, Boire G, van Schaardenburg D, Wichuk S, Turk S, Boers M, Siminovitch KA, Bykerk V, Keystone E, Tak PP, van Kuijk AW, Landewe R, van der Heijde D, Murphy M, Marotta A. 14-3-3eta Autoantibodies: Diagnostic Use in Early Rheumatoid Arthritis. J Rheumatol. 2015 Sep;42(9):1587-94. doi: 10.3899/jrheum.141385. Epub 2015 Jul 15. PMID 26178283
- [Background] Leblanc-Trudeau C, Dobkin PL, Carrier N, Cossette P, de Brum-Fernandes AJ, Liang P, Masetto A, Boire G. Depressive symptoms predict future simple disease activity index scores and simple disease activity index remission in a prospective cohort of patients with early inflammatory polyarthritis. Rheumatology (Oxford). 2015 Dec;54(12):2205-14. doi: 10.1093/rheumatology/kev272. Epub 2015 Jul 25. PMID 26209789
- [Background] Challener GJ, Jones JD, Pelzek AJ, Hamilton BJ, Boire G, de Brum-Fernandes AJ, Masetto A, Carrier N, Menard HA, Silverman GJ, Rigby WFC. Anti-carbamylated Protein Antibody Levels Correlate with Anti-Sa (Citrullinated Vimentin) Antibody Levels in Rheumatoid Arthritis. J Rheumatol. 2016 Feb;43(2):273-281. doi: 10.3899/jrheum.150179. Epub 2015 Dec 15. PMID 26669911
- [Background] Carrier N, Marotta A, de Brum-Fernandes AJ, Liang P, Masetto A, Menard HA, Maksymowych WP, Boire G. Serum levels of 14-3-3eta protein supplement C-reactive protein and rheumatoid arthritis-associated antibodies to predict clinical and radiographic outcomes in a prospective cohort of patients with recent-onset inflammatory polyarthritis. Arthritis Res Ther. 2016 Feb 1;18:37. doi: 10.1186/s13075-016-0935-z. PMID 26832367
- [Result] Boire G, Cossette P, de Brum-Fernandes AJ, Liang P, Niyonsenga T, Zhou ZJ, Carrier N, Daniel C, Menard HA. Anti-Sa antibodies and antibodies against cyclic citrullinated peptide are not equivalent as predictors of severe outcomes in patients with recent-onset polyarthritis. Arthritis Res Ther. 2005;7(3):R592-603. doi: 10.1186/ar1719. Epub 2005 Mar 17. PMID 15899046
- [Result] Guzian MC, Carrier N, Cossette P, de Brum-Fernandes AJ, Liang P, Menard HA, Boire G. Outcomes in recent-onset inflammatory polyarthritis differ according to initial titers, persistence over time, and specificity of the autoantibodies. Arthritis Care Res (Hoboken). 2010 Nov;62(11):1624-32. doi: 10.1002/acr.20288. Epub 2010 Jul 8. PMID 20617532
- [Result] Carrier N, Cossette P, Daniel C, de Brum-Fernandes A, Liang P, Menard HA, Boire G. The DERAA HLA-DR alleles in patients with early polyarthritis: protection against severe disease and lack of association with rheumatoid arthritis autoantibodies. Arthritis Rheum. 2009 Mar;60(3):698-707. doi: 10.1002/art.24353. PMID 19248090
- [Result] Dobkin PL, Liu A, Abrahamowicz M, Carrier N, de Brum-Fernandes AJ, Cossette P, Boire G. Predictors of pain for patients with early inflammatory polyarthritis. Arthritis Care Res (Hoboken). 2013 Jun;65(6):992-9. doi: 10.1002/acr.21923. PMID 23281243
- [Result] Maksymowych WP, van der Heijde D, Allaart CF, Landewe R, Boire G, Tak PP, Gui Y, Ghahary A, Kilani R, Marotta A. 14-3-3eta is a novel mediator associated with the pathogenesis of rheumatoid arthritis and joint damage. Arthritis Res Ther. 2014 Apr 21;16(2):R99. doi: 10.1186/ar4547. PMID 24751211
- [Result] Jones JD, Hamilton BJ, Challener GJ, de Brum-Fernandes AJ, Cossette P, Liang P, Masetto A, Menard HA, Carrier N, Boyle DL, Rosengren S, Boire G, Rigby WF. Serum C-X-C motif chemokine 13 is elevated in early and established rheumatoid arthritis and correlates with rheumatoid factor levels. Arthritis Res Ther. 2014 Apr 25;16(2):R103. doi: 10.1186/ar4552. PMID 24766912